CLINICAL TRIAL: NCT02484235
Title: Effects of High Intensity Interval Training, Strength Training and the Combination in Overweight and Obese
Brief Title: Effects of High Intensity Interval Training and Strength Training in Obese
Acronym: EHITSTR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Edgardo Opazo, PT, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: pro-001
Record Dates: First submitted 2015-06-23; First posted 2015-06-29 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Obesity
Keywords: obesity; exercise; HIIT; Vo2; kinetics
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group HIIT (Experimental): Only Aerobic Training with HIIT
  Interventions: Other: HIIT
- Group Strength (Experimental): Only Strength Training
  Interventions: Other: Strength
- HIIT and Strength (Experimental): Both intervention HIIT and Strength training
  Interventions: Other: HIIT; Other: Strength

INTERVENTIONS:
Other: HIIT — Group training with HIIT 3 times per week during 10 sessions
  Arms: Group HIIT; HIIT and Strength
Other: Strength — Group training with strength exercises 3 times per week during 10 sessions
  Arms: Group Strength; HIIT and Strength

SUMMARY:
Obesity is a global health problem since it is associated with many cardiovascular and metabolic diseases, osteoarticular problems and some cancers. That is why it is a priority of the national health policies. Exercise is a mainstay in the treatment, but still the most effective method is sought. The resistance exercise and high intensity intervals (HIIT) have been shown to positively affect the outcome of the disease, increasing the oxidative capacity of the trained subjects. Therefore it is important to look if both together produce greater benefits or otherwise nullify its effects, such as suggested by recent publications in relation to the cellular response to different stimuli such exercise in skeletal muscle. The aim of this study is to evaluate the effectiveness of interventions exercise high intensity intervals, overload and combining them in the oxidative capacity of obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Indication of medical supervised exercise
* BMI of 25-35kg/m2
* Participate in a 10 session rehabilitation program

Exclusion Criteria:

* Osteomuscular injuries
* Cardiovascular disease without control
* Bariatric Surgery
* High blood pressure without control

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Exercise Test of Vo2 kinetics | 6 weeks

SECONDARY OUTCOMES:
Strength test of 10 maximum repetition (10RM) | 6 weeks
Exercise test of max Walking Speed | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinico de la Universidad de Chile, Santiago, Santiago Metropolitan, Chile